CLINICAL TRIAL: NCT01897896
Title: An Open-Label, Long Term Safety Study of SD-809 ER in Subjects With Chorea Associated With Huntington Disease
Brief Title: Alternatives for Reducing Chorea in Huntington Disease
Acronym: ARC-HD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Auspex Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SD-809-C-16
Record Dates: First submitted 2013-06-14; First posted 2013-07-12 (Estimated); Results first posted 2019-04-16 (Actual); Last update posted 2021-11-09 (Actual); Status verified 2021-11

CONDITIONS: Chorea Associated With Huntington Disease
Keywords: Chorea; Huntington Disease
MeSH Terms: conditions — Chorea; Huntington Disease | interventions — deutetrabenazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Rollover Cohort: SD-809 ER (Experimental): Participants who completed study SD-809-C-15 (NCT01795859, including 1-week washout period and Week 13 evaluation), will receive 6 milligrams (mg) SD-809 ER tablet once daily as a starting dose in this study. Dose titration will be continued through Week 8 to optimize dose. Dose of SD-809 ER can be adjusted weekly in increments of 6 milligrams per day (mg/day) (6 or 12 mg/day after a total daily dose of 48 mg is reached) based on chorea control and adverse events. Daily doses of SD-809 ER 12 mg and higher will be administered twice daily. Maximum total daily dose of SD-809 ER will be 72 mg/day (36 mg twice daily), unless participant is receiving a strong CYP2D6 inhibitor(such as, paroxetine, buproprion, fluoxetine), in which case maximum total daily dose will be 42 mg (21 mg twice daily). Long-term treatment with SD-809 ER at a stable dose (further dose adjustments are permitted, if clinically indicated) will be continued until SD-809 ER become commercially available in United States.
  Interventions: Drug: SD-809
- Switch Cohort: SD-809 ER (Experimental): Participants who were receiving an approved dosing regimen of tetrabenazine for at least 8 weeks prior to screening, will be converted overnight from their existing tetrabenazine regimen to SD-809 ER regimen to achieve targeted steady-state area under the curve (AUC) of total (alpha+beta)- Dihydrotetrabenazine (HTBZ) metabolites that is predicted to be comparable to that of participant's prior tetrabenazine regimen. Participants will remain on initial dose of SD-809 ER through Week 1. Dose adjustment will be continued through Week 4 to optimize the dose. Dose of SD-809 ER can be adjusted weekly (upward or downward) in increments of 6 mg per day (6 mg/day or 12 mg/day after a total daily dose of 48 mg is reached), based on chorea control and treatment regimen tolerability. Long-term treatment with SD-809 ER at a stable dose (although further dose adjustments are permitted, if clinically indicated) will be continued until SD-809 ER become commercially available in United States.
  Interventions: Drug: SD-809

INTERVENTIONS:
Drug: SD-809 — SD-809 tablets will be provided in dose strengths of 6, 9 and 12 mg.
  Other Names: Deutetrabenazine

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and pharmacokinetics of SD-809 extended release (ER) in participants switching from tetrabenazine to SD-809 ER. In addition, the safety and tolerability of long-term treatment with SD-809 ER will be assessed in "Switch" participants as well as "Rollover" participants completing a randomized, double blind, placebo-controlled study of SD-809 ER.

ELIGIBILITY:
Inclusion Criteria:

* Participant is at least 18 years of age or the age of majority (whichever is older) at Screening.
* Participant has been diagnosed with manifest HD, as indicated by characteristic motor exam features, and has a documented expanded cytosine adenine guanine (CAG) repeat (greater than or equal to >= [37]) at or before Screening.
* Participant meets either of the following:

  1. Has successfully completed participation in the First-HD Study (SD-809-C-15) or
  2. Has been receiving an Food and Drug Administration (FDA)-approved dose of tetrabenazine that has been stable for >=8 weeks before Screening and is providing a therapeutic benefit for control of chorea.
* Participant has a Total Functional Capacity (TFC) score >=5 at Screening.
* Participant is able to swallow study medication whole.
* Participant has provided written, informed consent or, a legally authorized representative (LAR) has provided written informed consent and the subject has provided assent.
* Participant has provided a Research Advance Directive.
* Female participants of childbearing potential agree to use an acceptable method of contraception from screening through study completion.
* The participant has a reliable caregiver who interacts with the participant on a daily basis, oversees study drug administration, assures attendance at study visits and participates in evaluations, as required.
* Participant is able to ambulate without assistance for at least 20 yards (Note: The use of assistive devices (such as; walker, cane) are permitted during ambulation).
* Has sufficient reading skills to comprehend the participant completed rating scales.

Exclusion Criteria:

* Participant has a serious untreated or under-treated psychiatric illness, such as depression, at Screening or Baseline.
* Participant has active suicidal ideation at Screening or Baseline.
* Participant has history of suicidal behavior at Screening or Baseline.
* Participant has evidence for depression at Baseline.
* Participant has an unstable or serious medical illness at Screening or Baseline.
* Participant has received tetrabenazine within 7 days of Baseline (Rollover participants only).
* Participant has received any of the following concomitant medications within 30 days of Screening or Baseline: Antipsychotics, Metoclopramide, Monoamine oxidase inhibitors (MAOI), Levodopa or dopamine agonists, Reserpine, Amantadine, Memantine (Rollover participants only)
* Switch participants may receive Memantine if on a stable, approved dose for at least 30 days
* Participant has significantly impaired swallowing function at Screening or Baseline.
* Participant has significantly impaired speaking at Screening or Baseline.
* Participant requires treatment with drugs known to prolong the QT interval.
* Participant has prolonged QT interval on 12-lead electrocardiogram (ECG) at Screening.
* Participant has evidence of hepatic impairment at Screening.
* Participant has evidence of significant renal impairment at Screening.
* Participant has known allergy to any of the components of study medication.
* Participant has participated in an investigational drug or device trial other than SD-809-C-15 within 30 days (or 5 drug half-lives) of Screening, whichever is longer.
* Participant is pregnant or breast-feeding at Screening or Baseline.
* Participant acknowledges present use of illicit drugs at Screening or Baseline.
* Participant has a history of alcohol or substance abuse in the previous 12 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2013-11-12 (Actual); Primary Completion 2017-08-21 (Actual); Study Completion 2017-08-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Teva Medical Expert, MD, Study Director — Teva Branded Pharmaceutical Products R&D, Inc.
Locations (38):
- United States (34):
  - Teva Investigational Site 057, Birmingham, Alabama
  - Teva Investigational Site 038, Phoenix, Arizona
  - Teva Investigational Site 298, Fayetteville, Arkansas
  - Teva Investigational Site 052, Englewood, Colorado
  - Teva Investigational Site 333, Washington D.C., District of Columbia
  - Teva Investigational Site 160, Gainesville, Florida
  - Teva Investigational Site 014, Miami, Florida
  - Teva Investigational Site 032, Atlanta, Georgia
  - Teva Investigational Site 045, Indianapolis, Indiana
  - Teva Investigational Site 024, Iowa City, Iowa
  - Teva Investigational Site 029, Kansas City, Kansas
  - Teva Investigational Site 083, Wichita, Kansas
  - Teva Investigational Site 087, Louisville, Kentucky
  - Teva Investigational Site 028, Baltimore, Maryland
  - Teva Investigational Site 040, Boston, Massachusetts
  - Teva Investigational Site 027, St Louis, Missouri
  - Teva Investigational Site 194, Las Vegas, Nevada
  - Teva Investigational Site 328, Camden, New Jersey
  - Teva Investigational Site 026, New Brunswick, New Jersey
  - Teva Investigational Site 037, Albany, New York
  - Teva Investigational Site 002, New York, New York
  - Teva Investigational Site 342, Patchogue, New York
  - Teva Investigational Site 119, Durham, North Carolina
  - Teva Investigational Site 089, Cincinnati, Ohio
  - Teva Investigational Site 020, Columbus, Ohio
  - Teva Investigational Site 093, Toledo, Ohio
  - Teva Investigational Site 341, Tulsa, Oklahoma
  - Teva Investigational Site 031, Nashville, Tennessee
  - Teva Investigational Site 007, Houston, Texas
  - Teva Investigational Site 199, Houston, Texas
  - Teva Investigational Site 100, Salt Lake City, Utah
  - Teva Investigational Site 137, Burlington, Vermont
  - Teva Investigational Site 220, Kirkland, Washington
  - Teva Investigational Site 096, Seattle, Washington
- Teva Investigational Site 054, Sydney, Australia
- Canada (3):
  - Teva Investigational Site 098, Montreal
  - Teva Investigational Site 231, Ottawa
  - Teva Investigational Site 300, Toronto

REFERENCES:
- [Derived] Frank S, Testa CM, Goldstein J, Kayson E, Leavitt BR, Oakes D, O'Neill C, Whaley J, Gross N, Chaijale N, Barash S, Gordon MF; Huntington Study Group/ARC-HD Investigators and Coordinators. Safety and Efficacy of Deutetrabenazine at High versus Lower Daily Dosages in the ARC-HD Study to Treat Chorea in Huntington Disease. CNS Drugs. 2025 Feb;39(2):185-195. doi: 10.1007/s40263-024-01139-3. Epub 2025 Jan 18. PMID 39825184
- [Derived] Frank S, Anderson KE, Fernandez HH, Hauser RA, Claassen DO, Stamler D, Factor SA, Jimenez-Shahed J, Barkay H, Wilhelm A, Alexander JK, Chaijale N, Barash S, Savola JM, Gordon MF, Chen M. Safety of Deutetrabenazine for the Treatment of Tardive Dyskinesia and Chorea Associated with Huntington Disease. Neurol Ther. 2024 Jun;13(3):655-675. doi: 10.1007/s40120-024-00600-1. Epub 2024 Apr 1. PMID 38557959
- [Derived] Frank S, Testa C, Edmondson MC, Goldstein J, Kayson E, Leavitt BR, Oakes D, O'Neill C, Vaughan C, Whaley J, Gross N, Gordon MF, Savola JM; Huntington Study Group/ARC-HD Investigators and Coordinators. The Safety of Deutetrabenazine for Chorea in Huntington Disease: An Open-Label Extension Study. CNS Drugs. 2022 Nov;36(11):1207-1216. doi: 10.1007/s40263-022-00956-8. Epub 2022 Oct 15. PMID 36242718

RESULTS

PARTICIPANT FLOW:
Groups:
- Rollover Cohort: SD-809 ER: Participants who completed study SD-809-C-15 (either placebo or SD-809 group [NCT01795859], including 1-week washout period and Week 13 evaluation), received 6 milligrams(mg) SD-809 ER tablet once daily as starting dose in this study. Dose titration was continued through Week 8 to optimize dose. SD-809 ER dose could be adjusted weekly in increments of 6 milligrams per day(mg/day) (6 or 12 mg/day after total daily dose of 48 mg reached) based on chorea control and adverse events. Daily doses of SD-809 ER 12 mg and higher were administered twice daily. Maximum total daily dose of SD-809 ER was 72 mg/day(36 mg twice daily), unless participant was receiving a strong CYP2D6 inhibitor(e.g., paroxetine,buproprion, fluoxetine), in which case maximum total daily dose was 42 mg (21 mg twice daily). Long-term treatment with SD-809 ER at stable dose (although further dose adjustments were permitted, if clinically indicated) continued until SD-809 ER became commercially available in United States.
- Switch Cohort: SD-809 ER: Participants who were receiving Food and Drug Administration (FDA) - approved dosing regimen of tetrabenazine for at least 8 weeks prior to screening, were converted overnight from their existing tetrabenazine regimen to SD-809 ER regimen to achieve targeted steady-state area under the curve(AUC) of total (alpha+beta)-Dihydrotetrabenazine(HTBZ) metabolites that was predicted to be comparable to that of participant's prior tetrabenazine regimen. Participants remained on initial dose of SD-809 ER through Week 1. Dose adjustment was continued through Week 4 to optimize the dose. SD-809 ER dose could be adjusted weekly (upward or downward) in increments of 6 mg per day (6 mg/day or 12 mg/day after total daily dose of 48 mg reached), based on chorea control and treatment regimen tolerability. Long-term treatment with SD-809 ER at stable dose (although further dose adjustments were permitted, if clinically indicated) continued until SD-809 ER became commercially available in United States.
Period: Overall Study
Arm/Group | Rollover Cohort: SD-809 ER | Switch Cohort: SD-809 ER
Started | 82 | 37
Completed | 56 | 25
Not Completed | 26 | 12
Not completed — Death | 1 | 0
Not completed — Adverse Event | 11 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Non-compliance with study drug dosing | 1 | 1
Not completed — Withdrawal by Subject | 7 | 1
Not completed — Require drug that interfere with study | 1 | 4
Not completed — Protocol Violation | 1 | 1
Not completed — Withdrawal per Investigator's judgement | 1 | 1
Not completed — Caregiver can no longer participate | 0 | 2
Not completed — Other than specified | 2 | 1

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who were administered at least 1 dose of drug.
Groups:
- Rollover Cohort: SD-809 ER: Participants who completed study SD-809-C-15 (either placebo group or SD-809 group, including 1-week washout period and Week 13 evaluation), received 6 mg SD-809 ER tablet once daily as a starting dose in this study. Dose titration was continued through Week 8 to optimize the dose. Dose of SD-809 ER could be adjusted weekly in increments of 6 mg/day (6 or 12 mg/day after a total daily dose of 48 mg was reached) based on chorea control and adverse events. Daily doses of SD-809 ER 12 mg and higher were administered twice daily. Maximum total daily dose of SD-809 ER was 72 mg/day (36 mg twice daily), unless the participant was receiving a strong CYP2D6 inhibitor (e.g., paroxetine, buproprion, and fluoxetine), in which case the maximum total daily dose was 42 mg (21 mg twice daily). Long-term treatment with SD-809 ER at a stable dose (although further dose adjustments were permitted, if clinically indicated) continued until SD-809 ER became commercially available in United States.
- Switch Cohort: SD-809 ER: Participants who were receiving FDA-approved dosing regimen of tetrabenazine for at least 8 weeks prior to screening, were converted overnight from their existing tetrabenazine regimen to SD-809 ER regimen to achieve targeted steady-state AUC of total (alpha+beta)-HTBZ metabolites that was predicted to be comparable to that of participant's prior tetrabenazine regimen. Participants remained on initial dose of SD-809 ER through Week 1. Dose adjustment was continued through Week 4 to optimize the dose. Dose of SD-809 ER could be adjusted weekly (upward or downward) in increments of 6 mg per day (6 mg/day or 12 mg/day after a total daily dose of 48 mg was reached), based on chorea control and treatment regimen tolerability. Long-term treatment with SD-809 ER at a stable dose (although further dose adjustments were permitted, if clinically indicated) continued until SD-809 ER became commercially available in United States.
- Total: Total of all reporting groups
Arm/Group | Rollover Cohort: SD-809 ER | Switch Cohort: SD-809 ER | Total
Number analyzed (Participants) | 82 | 37 | 119
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.7 (12.27) | 52.4 (11.48) | 53.3 (12.00)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 15 | 52
  Male | 45 | 22 | 67
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 82 | 35 | 117
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 4 | 0 | 4
  White | 76 | 36 | 112
  Other | 0 | 1 | 1
  Multiple | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs), Serious TEAEs, Severe TEAEs, Drug-Related TEAEs, and TEAEs Leading to Withdrawal During Entire Treatment Period
Description: An adverse event (AE) was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Severe AE=inability to carry out usual activities. Drug-related TEAEs: TEAEs with possible, probable, definite, or missing relationship to study drug. Serious AEs: death, a life-threatening AE, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, a congenital anomaly or birth defect, or an important medical event that jeopardized participant and required medical intervention to prevent 1 of the outcomes listed in this definition. TEAEs: events that 1) began after treatment with study drug in current study and that were not present at baseline or 2) if present at baseline, had worsened in severity. Any TEAEs included both serious and non-serious TEAEs. A summary of other non-serious AEs and all serious AEs, regardless of causality is located in Reported AE section.
Time Frame: Baseline to follow-up visit (up to approximately 3 years 9 months)
Population: Safety population included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Rollover Cohort: SD-809 ER | Switch Cohort: SD-809 ER
Number analyzed (Participants) | 82 | 37
Participants
  Any TEAEs | 77 | 35
  Serious TEAEs | 21 | 11
  Severe TEAEs | 17 | 7
  Drug-Related TEAEs | 56 | 26
  TEAEs Leading to Withdrawal From Study | 13 | 3

2. Primary Outcome: Rollover Cohort: Number of Participants With TEAEs, Serious TEAEs, Severe TEAEs, Drug-Related TEAEs, and TEAEs Leading to Withdrawal During Titration
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Severe AEs=inability to carry out usual activities. Drug-related TEAEs: TEAEs with a possible, probable, definite, or missing relationship to study drug. Serious AEs: death, a life-threatening AE, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, a congenital anomaly or birth defect, or an important medical event that jeopardized the participant and required medical intervention to prevent 1 of the outcomes listed in this definition. TEAEs: events that 1) began after treatment with study drug in current study and that were not present at baseline or 2) if present at baseline, had worsened in severity. Any TEAEs included both serious and non-serious TEAEs. A summary of other non-serious AEs and all serious AEs, regardless of causality is located in Reported AE section.
Time Frame: Day 1 to end of Week 8
Population: Safety population included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Rollover Cohort: SD-809 ER
Number analyzed (Participants) | 82
Participants
  Any TEAEs | 49
  Serious TEAEs | 1
  Severe TEAEs | 0
  Drug-Related TEAEs | 23
  TEAEs Leading to Withdrawal From Study | 0

3. Primary Outcome: Switch Cohort: Number of Participants With TEAEs, Serious TEAEs, Severe TEAEs, Drug-Related TEAEs, and TEAEs Leading to Withdrawal During Dose Adjustment
Description: as for outcome 2
Time Frame: Day 1 to end of Week 4
Population: Safety population included all participants received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Switch Cohort: SD-809 ER
Number analyzed (Participants) | 37
Participants
  Any TEAEs | 17
  Serious TEAEs | 1
  Severe TEAEs | 1
  Drug-Related TEAEs | 11
  TEAEs Leading to Withdrawal From Study | 0

4. Primary Outcome: Number of Participants With TEAEs, Serious TEAEs, Severe TEAEs, Drug-Related TEAEs, and TEAEs Leading to Withdrawal During Long Term Stable Dose Treatment
Description: as for outcome 2
Time Frame: Week 8 to follow-up visit (up to approximately 3 years 9 months)
Population: Safety population included all participants who received at least 1 dose of study drug. Here, 'Overall number of participants analyzed' signifies number of participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Rollover Cohort: SD-809 ER | Switch Cohort: SD-809 ER
Number analyzed (Participants) | 81 | 35
Participants
  Any TEAEs | 74 | 35
  Serious TEAEs | 20 | 10
  Severe TEAEs | 17 | 7
  Drug-Related TEAEs | 49 | 22
  TEAEs Leading to Withdrawal From Study | 13 | 3

5. Secondary Outcome: Change From Baseline in Clinical Laboratory Hematology Parameters (Basophils, Eosinophils, Leukocytes, Lymphocytes, Monocytes, Neutrophils and Platelets) at Week 158
Description: Clinical laboratory hematology parameters included basophils, eosinophils, leukocytes, lymphocytes, monocytes, neutrophils, platelets, erythrocytes mean corpuscular volume, erythrocytes, hematocrit, and hemoglobin. Change from baseline in basophils, eosinophils, leukocytes, lymphocytes, monocytes, neutrophils and platelets cells at baseline and Week 158 is reported in this outcome measure. Observed value at baseline and observed values at Week 158 were used to calculate the change from baseline value at Week 158.
Time Frame: Baseline, Week 158
Population: Safety population included all participants who received at least 1 dose of study drug. Here, 'Number analyzed' signifies participants evaluable for this outcome measure for specified categories.
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter
Arm/Group | Rollover Cohort: SD-809 ER | Switch Cohort: SD-809 ER
Number analyzed (Participants) | 82 | 37
10^9 cells per liter
  Basophils: Baseline | 0.029 (0.0231) | 0.035 (0.0283)
  Basophils: Change at Week 158: number analyzed (Participants) | 18 | 8
  Basophils: Change at Week 158 | -0.014 (0.0287) | -0.004 (0.0385)
  Eosinophils: Baseline | 0.151 (0.1274) | 0.195 (0.1366)
  Eosinophils: Change at Week 158: number analyzed (Participants) | 18 | 8
  Eosinophils: Change at Week 158 | -0.054 (0.0784) | 0.009 (0.0911)
  Leukocytes: Baseline | 6.98 (2.083) | 6.97 (1.828)
  Leukocytes: Change at Week 158: number analyzed (Participants) | 18 | 8
  Leukocytes: Change at Week 158 | -0.04 (0.927) | -0.04 (1.098)
  Lymphocytes: Baseline | 1.922 (0.7674) | 1.789 (0.7088)
  Lymphocytes: Change at Week 158: number analyzed (Participants) | 18 | 8
  Lymphocytes: Change at Week 158 | -0.088 (0.4261) | 0.075 (0.5409)
  Monocytes: Baseline | 0.445 (0.1805) | 0.416 (0.1416)
  Monocytes: Change at Week 158: number analyzed (Participants) | 18 | 8
  Monocytes: Change at Week 158 | -0.129 (0.1722) | -0.068 (0.1335)
  Neutrophils: Baseline | 4.437 (1.6324) | 4.538 (1.4741)
  Neutrophils: Change at Week 158: number analyzed (Participants) | 18 | 8
  Neutrophils: Change at Week 158 | 0.243 (0.6359) | -0.050 (0.8166)
  Platelets: Baseline | 235.6 (62.81) | 247.2 (77.63)
  Platelets: Change at Week 158: number analyzed (Participants) | 18 | 8
  Platelets: Change at Week 158 | 1.2 (56.09) | -12.0 (26.59)

6. Secondary Outcome: Change From Baseline in Clinical Laboratory Hematology Parameter (Erythrocytes Mean Corpuscular Volume) at Week 158
Description: Clinical laboratory hematology parameters included basophils, eosinophils, leukocytes, lymphocytes, monocytes, neutrophils, platelets, erythrocytes mean corpuscular volume, erythrocytes, hematocrit, and hemoglobin. Change from baseline in erythrocytes mean corpuscular volume at baseline and Week 158 is reported in this outcome measure. Observed value at baseline and observed value at Week 158 were used to calculate the change from baseline value at Week 158.
Time Frame: Baseline, Week 158
Population: Safety population included all participants received at least 1 dose of study drug. Here, 'Number analyzed' signifies participants evaluable for this outcome measure at specified timepoints.
Measure: Mean (Standard Deviation); unit: femtoliter (fL)
Arm/Group | Rollover Cohort: SD-809 ER | Switch Cohort: SD-809 ER
Number analyzed (Participants) | 82 | 37
femtoliter (fL)
  Baseline | 91.1 (3.95) | 92.1 (5.39)
  Change at Week 158: number analyzed (Participants) | 18 | 8
  Change at Week 158 | 2.2 (3.23) | 1.6 (4.14)

7. Secondary Outcome: Change From Baseline in Clinical Laboratory Hematology Parameter (Erythrocytes) at Week 158
Description: Clinical laboratory hematology parameters included basophils, eosinophils, leukocytes, lymphocytes, monocytes, neutrophils, platelets, erythrocytes mean corpuscular volume, erythrocytes, hematocrit, and hemoglobin. Change from baseline in erythrocytes at baseline and Week 158 is reported in this outcome measure. Observed value at baseline and observed value at Week 158 were used to calculate the change from baseline value at Week 158.
Time Frame: Baseline, Week 158
Population: Safety population included all participants who received at least 1 dose of study drug. Here, 'Number analyzed' signifies participants evaluable for this outcome measure at specified timepoints.
Measure: Mean (Standard Deviation); unit: 10^12 cells per liter
Arm/Group | Rollover Cohort: SD-809 ER | Switch Cohort: SD-809 ER
Number analyzed (Participants) | 82 | 37
10^12 cells per liter
  Baseline | 4.60 (0.397) | 4.54 (0.377)
  Change at Week 158: number analyzed (Participants) | 18 | 8
  Change at Week 158 | 0.18 (0.262) | 0.19 (0.247)

8. Secondary Outcome: Change From Baseline in Clinical Laboratory Hematology Parameter (Hematocrit) at Week 158
Description: Clinical laboratory hematology parameters included basophils, eosinophils, leukocytes, lymphocytes, monocytes, neutrophils, platelets, erythrocytes mean corpuscular volume, erythrocytes, hematocrit, and hemoglobin. Hematocrit levels were calculated as the ratio of the volume of red cells to the volume of whole blood. Change from baseline in hematocrit at baseline and Week 158 is reported in this outcome measure. Observed value at baseline and observed value at Week 158 were used to calculate the change from baseline value at Week 158.
Time Frame: Baseline, Week 158
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Rollover Cohort: SD-809 ER | Switch Cohort: SD-809 ER
Number analyzed (Participants) | 82 | 37
ratio
  Baseline | 0.419 (0.0363) | 0.417 (0.0397)
  Change at Week 158: number analyzed (Participants) | 18 | 8
  Change at Week 158 | 0.025 (0.0255) | 0.025 (0.0334)

9. Secondary Outcome: Change From Baseline in Clinical Laboratory Hematology Parameter (Hemoglobin) at Week 158
Description: Clinical laboratory hematology parameters included basophils, eosinophils, leukocytes, lymphocytes, monocytes, neutrophils, platelets, erythrocytes mean corpuscular volume, erythrocytes, hematocrit, and hemoglobin. Change from baseline in hemoglobin at baseline and Week 158 is reported in this outcome measure. Observed value at baseline and observed value at Week 158 were used to calculate the change from baseline value at Week 158.
Time Frame: Baseline, Week 158
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: grams per liter (g/L)
Arm/Group | Rollover Cohort: SD-809 ER | Switch Cohort: SD-809 ER
Number analyzed (Participants) | 82 | 37
grams per liter (g/L)
  Baseline | 139.7 (12.26) | 138.4 (13.19)
  Change at Week 158: number analyzed (Participants) | 18 | 8
  Change at Week 158 | 4.6 (7.99) | 4.5 (11.99)

10. Secondary Outcome: Change From Baseline in Clinical Laboratory Serum Chemistry Parameters (Alanine Aminotransferase and Alkaline Phosphatase) at Week 158
Description: Clinical laboratory serum chemistry parameters included alanine aminotransferase, alkaline phosphatase, aspartate aminotransferase, lactate dehydrogenase, bicarbonate, blood urea nitrogen, calcium, chloride, cholesterol, glucose, magnesium, phosphate, potassium, sodium, triglycerides, protein, albumin, creatinine clearance, bilirubin, creatinine, direct bilirubin, and urate. Change from baseline in alanine aminotransferase and alkaline phosphatase at baseline and Week 158 is reported in this outcome measure. Observed value at baseline and observed value at Week 158 were used to calculate the change from baseline value at Week 158.
Time Frame: Baseline, Week 158
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: international units per liter (IU/L)
Arm/Group | Rollover Cohort: SD-809 ER | Switch Cohort: SD-809 ER
Number analyzed (Participants) | 82 | 37
international units per liter (IU/L)
  Alanine Aminotransferase: Baseline | 20.7 (9.74) | 18.9 (12.20)
  Alanine Aminotransferase: Change at Week 158: number analyzed (Participants) | 19 | 9
  Alanine Aminotransferase: Change at Week 158 | -5.3 (7.51) | -2.1 (9.74)
  Alkaline Phosphatase: Baseline | 72.6 (20.24) | 73.1 (20.61)
  Alkaline Phosphatase: Change at Week 158: number analyzed (Participants) | 19 | 9
  Alkaline Phosphatase: Change at Week 158 | -1.0 (8.21) | 1.0 (9.62)

11. Secondary Outcome: Change From Baseline in Clinical Laboratory Serum Chemistry Parameters (Aspartate Aminotransferase and Lactate Dehydrogenase) at Week 158
Description: Clinical laboratory serum chemistry parameters included alanine aminotransferase, alkaline phosphatase, aspartate aminotransferase, lactate dehydrogenase, bicarbonate, blood urea nitrogen, calcium, chloride, cholesterol, glucose, magnesium, phosphate, potassium, sodium, triglycerides, protein, albumin, creatinine clearance, bilirubin, creatinine, direct bilirubin, and urate. Change from baseline in aspartate aminotransferase and lactate dehydrogenase at baseline and Week 158 is reported in this outcome measure. Observed value at baseline and observed value at Week 158 were used to calculate the change from baseline value at Week 158.
Time Frame: Baseline, Week 158
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units per liter (U/L)
Arm/Group | Rollover Cohort: SD-809 ER | Switch Cohort: SD-809 ER
Number analyzed (Participants) | 82 | 37
units per liter (U/L)
  Aspartate Aminotransferase: Baseline | 20.5 (5.84) | 18.4 (6.88)
  Aspartate Aminotransferase: Change at Week 158: number analyzed (Participants) | 19 | 9
  Aspartate Aminotransferase: Change at Week 158 | -2.7 (5.43) | -1.1 (5.40)
  Lactate Dehydrogenase: Baseline: number analyzed (Participants) | 81 | 37
  Lactate Dehydrogenase: Baseline | 163.9 (28.05) | 161.1 (42.32)
  Lactate Dehydrogenase: Change at Week 158: number analyzed (Participants) | 19 | 9
  Lactate Dehydrogenase: Change at Week 158 | -5.5 (27.83) | -4.9 (18.45)

12. Secondary Outcome: Change From Baseline in Clinical Laboratory Serum Chemistry Parameters (Bicarbonate, Blood Urea Nitrogen, Calcium, Chloride, Cholesterol, Glucose, Magnesium, Phosphate, Potassium, Sodium, Triglycerides) at Week 158
Description: Clinical laboratory serum chemistry parameters included alanine aminotransferase, alkaline phosphatase, aspartate aminotransferase, lactate dehydrogenase, bicarbonate, blood urea nitrogen, calcium, chloride, cholesterol, glucose, magnesium, phosphate, potassium, sodium, triglycerides, protein, albumin, creatinine clearance, bilirubin, creatinine, direct bilirubin, and urate. Change from baseline in bicarbonate, blood urea nitrogen, calcium, chloride, cholesterol, glucose, magnesium, phosphate, potassium, sodium and triglycerides at baseline and Week 158 is reported in this outcome measure. Observed value at baseline and observed value at Week 158 were used to calculate the change from baseline value at Week 158.
Time Frame: Baseline, Week 158
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: millimoles per liter (mmol/L)
Arm/Group | Rollover Cohort: SD-809 ER | Switch Cohort: SD-809 ER
Number analyzed (Participants) | 82 | 37
millimoles per liter (mmol/L)
  Bicarbonate: Baseline | 24.7 (2.55) | 24.7 (2.06)
  Bicarbonate: Change at Week 158: number analyzed (Participants) | 19 | 9
  Bicarbonate: Change at Week 158 | -0.2 (2.87) | 0.7 (3.16)
  Blood Urea Nitrogen: Baseline | 5.979 (1.8432) | 6.282 (1.8177)
  Blood Urea Nitrogen: Change at Week 158: number analyzed (Participants) | 19 | 9
  Blood Urea Nitrogen: Change at Week 158 | -0.531 (1.4864) | -0.323 (0.9797)
  Calcium: Baseline | 2.417 (0.1067) | 2.393 (0.1523)
  Calcium: Change at Week 158: number analyzed (Participants) | 19 | 9
  Calcium: Change at Week 158 | -0.034 (0.1282) | -0.067 (0.0869)
  Chloride: Baseline | 102.5 (2.28) | 103.8 (2.24)
  Chloride: Change at Week 158: number analyzed (Participants) | 19 | 9
  Chloride: Change at Week 158 | -2.7 (2.62) | -2.0 (1.50)
  Cholesterol: Baseline | 5.118 (0.9505) | 4.863 (1.1686)
  Cholesterol: Change at Week 158: number analyzed (Participants) | 19 | 9
  Cholesterol: Change at Week 158 | -0.131 (0.8790) | -0.173 (0.7715)
  Glucose: Baseline | 5.28 (1.571) | 5.31 (1.029)
  Glucose: Change at Week 158: number analyzed (Participants) | 19 | 9
  Glucose: Change at Week 158 | -0.54 (1.018) | -0.64 (1.033)
  Magnesium: Baseline | 0.871 (0.0566) | 0.843 (0.0567)
  Magnesium: Change at Week 158: number analyzed (Participants) | 19 | 9
  Magnesium: Change at Week 158 | -0.027 (0.0701) | 0.016 (0.0639)
  Phosphate: Baseline | 1.194 (0.1769) | 1.191 (0.1661)
  Phosphate: Change at Week 158: number analyzed (Participants) | 19 | 9
  Phosphate: Change at Week 158 | -0.029 (0.2298) | 0.061 (0.1330)
  Potassium: Baseline | 4.39 (0.419) | 4.46 (0.332)
  Potassium: Change at Week 158: number analyzed (Participants) | 19 | 9
  Potassium: Change at Week 158 | -0.14 (0.414) | 0.19 (0.501)
  Sodium: Baseline | 142.4 (2.14) | 142.9 (2.31)
  Sodium: Change at Week 158: number analyzed (Participants) | 19 | 9
  Sodium: Change at Week 158 | -2.0 (3.56) | -1.7 (2.06)
  Triglycerides: Baseline | 1.606 (1.0001) | 1.733 (1.2887)
  Triglycerides: Change at Week 158: number analyzed (Participants) | 19 | 9
  Triglycerides: Change at Week 158 | -0.147 (0.8692) | -0.420 (1.0005)

13. Secondary Outcome: Change From Baseline in Clinical Laboratory Serum Chemistry Parameters (Protein and Albumin) at Week 158
Description: Clinical laboratory serum chemistry parameters included alanine aminotransferase, alkaline phosphatase, aspartate aminotransferase, lactate dehydrogenase, bicarbonate, blood urea nitrogen, calcium, chloride, cholesterol, glucose, magnesium, phosphate, potassium, sodium, triglycerides, protein, albumin, creatinine clearance, bilirubin, creatinine, direct bilirubin, and urate. Change from baseline in protein and albumin at baseline and Week 158 is reported in this outcome measure. Observed value at baseline and observed value at Week 158 were used to calculate the change from baseline value at Week 158.
Time Frame: Baseline, Week 158
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Rollover Cohort: SD-809 ER | Switch Cohort: SD-809 ER
Number analyzed (Participants) | 82 | 37
g/L
  Protein: Baseline | 69.5 (3.88) | 67.3 (4.54)
  Protein: Change at Week 158: number analyzed (Participants) | 19 | 9
  Protein: Change at Week 158 | -0.9 (3.54) | -2.9 (4.43)
  Albumin: Baseline | 43.9 (2.55) | 43.1 (2.65)
  Albumin: Change at Week 158: number analyzed (Participants) | 19 | 9
  Albumin: Change at Week 158 | 0.2 (3.61) | -0.9 (2.57)

14. Secondary Outcome: Change From Baseline in Clinical Laboratory Serum Chemistry Parameter (Creatinine Clearance) at Week 106
Description: Clinical laboratory serum chemistry parameters included alanine aminotransferase, alkaline phosphatase, aspartate aminotransferase, lactate dehydrogenase, bicarbonate, blood urea nitrogen, calcium, chloride, cholesterol, glucose, magnesium, phosphate, potassium, sodium, triglycerides, protein, albumin, creatinine clearance, bilirubin, creatinine, direct bilirubin, and urate. Change from baseline in creatinine clearance at baseline and Week 106 is reported in this outcome measure. Observed value at baseline and observed value at Week 106 were used to calculate the change from baseline value at Week 106.
Time Frame: Baseline, Week 106
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: milliliters per minute (mL/min)
Arm/Group | Rollover Cohort: SD-809 ER | Switch Cohort: SD-809 ER
Number analyzed (Participants) | 82 | 37
milliliters per minute (mL/min)
  Baseline: number analyzed (Participants) | 81 | 36
  Baseline | 94.1 (26.67) | 89.9 (27.55)
  Change at Week 106: number analyzed (Participants) | 2 | 1
  Change at Week 106 | -4.5 (6.36) | -34.0

15. Secondary Outcome: Change From Baseline in Clinical Laboratory Serum Chemistry Parameters (Bilirubin, Creatinine, Direct Bilirubin, and Urate) at Week 158
Description: Clinical laboratory serum chemistry parameters included alanine aminotransferase, alkaline phosphatase, aspartate aminotransferase, lactate dehydrogenase, bicarbonate, blood urea nitrogen, calcium, chloride, cholesterol, glucose, magnesium, phosphate, potassium, sodium, triglycerides, protein, albumin, creatinine clearance, bilirubin, creatinine, direct bilirubin, and urate. Change from baseline in bilirubin, creatinine, direct bilirubin, and urate at baseline and Week 158 is reported in this outcome measure. Observed value at baseline and observed value at Week 158 were used to calculate the change from baseline value at Week 158.
Time Frame: Baseline, Week 158
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: micromoles per liter
Arm/Group | Rollover Cohort: SD-809 ER | Switch Cohort: SD-809 ER
Number analyzed (Participants) | 82 | 37
micromoles per liter
  Bilirubin: Baseline | 7.8 (4.82) | 6.0 (2.43)
  Bilirubin: Change at Week 158: number analyzed (Participants) | 19 | 9
  Bilirubin: Change at Week 158 | -0.7 (2.51) | -1.4 (2.07)
  Creatinine: Baseline | 82.8 (16.81) | 84.2 (19.02)
  Creatinine: Change at Week 158: number analyzed (Participants) | 19 | 9
  Creatinine: Change at Week 158 | -2.4 (10.13) | -2.4 (6.46)
  Direct Bilirubin: Baseline: number analyzed (Participants) | 81 | 37
  Direct Bilirubin: Baseline | 2.4 (0.94) | 2.1 (0.35)
  Direct Bilirubin: Change at Week 158: number analyzed (Participants) | 19 | 9
  Direct Bilirubin: Change at Week 158 | 0.1 (0.23) | -0.2 (0.44)
  Urate: Baseline | 305.2 (83.70) | 269.5 (75.06)
  Urate: Change at Week 158: number analyzed (Participants) | 19 | 9
  Urate: Change at Week 158 | -21.8 (55.50) | -3.4 (39.37)

16. Secondary Outcome: Change From Baseline in Blood Pressure at Week 171
Description: Systolic blood pressure (SBP) and diastolic blood pressure (DBP) were assessed in seated/supine position. Observed value at baseline and observed value at Week 171 were used to calculate the change from baseline value at Week 171.
Time Frame: Baseline, Week 171
Population: Safety population included all participants who received at least 1 dose of study drug. Here, 'Number of participants analyzed' signifies participants evaluable for this outcome measure for specified categories.
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | Rollover Cohort: SD-809 ER | Switch Cohort: SD-809 ER
Number analyzed (Participants) | 82 | 37
millimeters of mercury (mmHg)
  SBP: Baseline: number analyzed (Participants) | 78 | 37
  SBP: Baseline | 120.5 (12.70) | 118.9 (17.80)
  SBP: Change at Week 171: number analyzed (Participants) | 1 | 0
  SBP: Change at Week 171 | -4.0 |
  DBP: Baseline: number analyzed (Participants) | 78 | 37
  DBP: Baseline | 73.3 (10.21) | 73.8 (11.85)
  DBP: Change at Week 171: number analyzed (Participants) | 1 | 0
  DBP: Change at Week 171 | -6.0 |

17. Secondary Outcome: Change From Baseline in Heart Rate at Week 171
Description: Heart rate was assessed in seated/supine position. Observed value at baseline and observed value at Week 171 were used to calculate the change from baseline value at Week 171.
Time Frame: Baseline, Week 171
Population: Safety population included all participants who received at least 1 dose of study drug. Here, 'Number of participants analyzed' signifies participants evaluable for this outcome measure at specified timepoints.
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Rollover Cohort: SD-809 ER | Switch Cohort: SD-809 ER
Number analyzed (Participants) | 82 | 37
beats per minute
  Baseline: number analyzed (Participants) | 78 | 37
  Baseline | 70.7 (8.68) | 68.1 (12.56)
  Change at Week 171: number analyzed (Participants) | 1 | 0
  Change at Week 171 | 25.0 |

18. Secondary Outcome: Change From Baseline in Respiration Rate at Week 171
Description: Observed value at baseline and observed value at Week 171 were used to calculate the change from baseline value at Week 171.
Time Frame: Baseline, Week 171
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: breaths/minute
Arm/Group | Rollover Cohort: SD-809 ER | Switch Cohort: SD-809 ER
Number analyzed (Participants) | 82 | 37
breaths/minute
  Baseline: number analyzed (Participants) | 78 | 37
  Baseline | 16.4 (2.57) | 17.5 (2.58)
  Change at Week 171: number analyzed (Participants) | 7 | 2
  Change at Week 171 | -1.3 (2.06) | -3.5 (3.54)

19. Secondary Outcome: Change From Baseline in Body Temperature at Week 171
Description: as for outcome 18
Time Frame: Baseline, Week 171
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: degrees centigrade
Arm/Group | Rollover Cohort: SD-809 ER | Switch Cohort: SD-809 ER
Number analyzed (Participants) | 82 | 37
degrees centigrade
  Baseline: number analyzed (Participants) | 79 | 37
  Baseline | 36.56 (0.427) | 36.67 (0.309)
  Change at Week 171: number analyzed (Participants) | 7 | 2
  Change at Week 171 | -0.13 (0.468) | -0.10 (0.283)

20. Secondary Outcome: Electrocardiogram (ECG) Parameter Value (Heart Rate) at Baseline and Week 8
Description: ECG parameters included heart rate, PR interval, QRS duration, QT interval and Fridericia's corrected QT interval (QTcF). Heart rate measured by ECG at Baseline and Week 8 is reported in this outcome measure.
Time Frame: Baseline, Week 8
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: beats/minute
Arm/Group | Rollover Cohort: SD-809 ER | Switch Cohort: SD-809 ER
Number analyzed (Participants) | 82 | 37
beats/minute
  Baseline | 67.4 (9.87) | 63.8 (13.96)
  Week 8: number analyzed (Participants) | 78 | 35
  Week 8 | 64.6 (9.22) | 65.8 (13.50)

21. Secondary Outcome: ECG Parameter Value (PR Interval, QRS Duration, QT Interval, QTcF) at Baseline and Week 8
Description: ECG parameters included heart rate, PR interval, QRS duration, QT interval and QTcF. PR interval, QRS duration, QT interval and QTcF at Baseline and Week 8 is reported in this outcome measure.
Time Frame: Baseline, Week 8
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Rollover Cohort: SD-809 ER | Switch Cohort: SD-809 ER
Number analyzed (Participants) | 82 | 37
milliseconds
  PR Interval: Baseline: number analyzed (Participants) | 81 | 37
  PR Interval: Baseline | 164.1 (25.03) | 159.5 (22.65)
  PR Interval: Week 8: number analyzed (Participants) | 78 | 35
  PR Interval: Week 8 | 165.2 (23.87) | 155.7 (18.08)
  QRS Duration: Baseline | 92.8 (14.37) | 88.8 (10.16)
  QRS Duration: Week 8: number analyzed (Participants) | 78 | 35
  QRS Duration: Week 8 | 91.0 (12.09) | 88.0 (10.97)
  QT Interval: Baseline | 399.8 (27.44) | 415.6 (37.44)
  QT Interval: Week 8: number analyzed (Participants) | 78 | 35
  QT Interval: Week 8 | 405.1 (29.10) | 404.5 (35.43)
  QTcF: Baseline | 413.3 (18.67) | 419.3 (17.89)
  QTcF: Week 8: number analyzed (Participants) | 78 | 35
  QTcF: Week 8 | 412.7 (20.10) | 412.8 (18.05)

22. Secondary Outcome: Number of Participants With Clinically Significant Abnormalities in ECG Parameters
Description: ECG parameters included heart rate, PR interval, QRS duration, QT interval and QTcF. Clinical significance was as as per Investigator's discretion.
Time Frame: Baseline, Week 8
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | Rollover Cohort: SD-809 ER | Switch Cohort: SD-809 ER
Number analyzed (Participants) | 82 | 37
Participants
  Baseline | 5 | 0
  Week 8: number analyzed (Participants) | 78 | 35
  Week 8 | 2 | 0

23. Secondary Outcome: Duration of Time to Achieve a Stable Dose of SD-809 ER
Description: Duration of time to achieve stable dose of SD-809, defined as the number of days from Day 1 until the first day at which the participant was taking the dose level they were receiving at Week 8.
Time Frame: From Day 1 until the first day at which the participant was taking the dose level they were receiving at Week 8 (up to maximum 1284 days)
Population: Safety population included all participants who received at least 1 dose of study drug. Here, 'Overall number of participants analyzed' signifies participants evaluable for this outcome measure.
Measure: Median (Full Range); unit: days
Arm/Group | Rollover Cohort: SD-809 ER | Switch Cohort: SD-809 ER
Number analyzed (Participants) | 81 | 35
days | 47.0 [1 to 73] | 28.0 [1 to 76]

24. Secondary Outcome: Change From Baseline in Unified Parkinson's Disease Rating Scale (UPDRS) -Dysarthria Score at Week 171
Description: The UPDRS is a comprehensive instrument used to assess the signs and symptoms of Parkinson's disease and includes patient and clinician-based assessments of motor, cognitive, and behavioral symptoms. The UPDRS-Dysarthria question pertaining to speech/dysarthria was used to monitor study participants for parkinsonism. Participants rated their responses on a scale ranging from 0 to 4, where 0 = normal; 1 = mildly affected, no difficulty being understood; 2 = moderately affected, sometimes asked to repeat statements; 3 = severely affected, frequently asked to repeat statements; 4 = unintelligible most of the time. Higher scores indicated greater impairment.
Time Frame: Baseline, Week 171
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rollover Cohort: SD-809 ER | Switch Cohort: SD-809 ER
Number analyzed (Participants) | 82 | 37
units on a scale
  Baseline: number analyzed (Participants) | 78 | 37
  Baseline | 0.9 (0.79) | 1.1 (0.74)
  Change at Week 171: number analyzed (Participants) | 7 | 2
  Change at Week 171 | 0.4 (0.79) | 1.5 (0.71)

25. Secondary Outcome: Change From Baseline in Barnes Akathisia Rating Scale (BARS) Summary Score at Week 171
Description: BARS is a rating scale for evaluation of drug-induced akathisia. It includes a summary score (objective assessment of akathisia and subjective measures [self-awareness and distress]) and a global clinical assessment. Objective akathisia rated on a scale of 0-3 (0=normal, occasional fidgety movements of limbs; 1=characteristic restless movements for less than half the time observed; 2= characteristic restless movements for at least half the time observed; 3=constant characteristic restless movements). Subjective measures included awareness of restlessness (rated on a scale of 0 [absence of inner restlessness] to 3 [awareness of intense compulsion to move]) and distress related to restlessness (rated on a scale of 0 [no distress] to 3 [severe distress]). Objective akathisia and subjective measures summed to yield summary score ranging from 0 (no akathisia and restlessness) to 9 (severe akathisia and restlessness), where higher scores indicated more akathisia and restlessness.
Time Frame: Baseline, Week 171
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rollover Cohort: SD-809 ER | Switch Cohort: SD-809 ER
Number analyzed (Participants) | 82 | 37
units on a scale
  Baseline: number analyzed (Participants) | 78 | 37
  Baseline | 1.1 (1.67) | 0.8 (1.25)
  Change at Week 171: number analyzed (Participants) | 7 | 2
  Change at Week 171 | 0.7 (1.50) | 0.5 (3.54)

26. Secondary Outcome: Change From Baseline in Barnes Akathisia Rating Scale (BARS) Global Assessment Score at Week 171
Description: BARS is a rating scale for evaluation of drug-induced akathisia. It includes a summary score (objective assessment of akathisia and subjective measures [self-awareness and distress]) and a global clinical assessment. Global clinical assessment rated on a scale ranging from 0 to 5, where 0=Absent. No evidence of awareness of restlessness; 1=Questionable. Non-specific inner tension and fidgety movements; 2=Mild akathisia. Awareness of restlessness in legs and/or inner restlessness worse when required to stand still. Fidgety movements present, but characteristic restless movements not necessarily observed; 3=Moderate akathisia. Awareness of restlessness combined with characteristic restless movements; 4=Marked akathisia. Subjective experience of restlessness includes a compulsive desire to walk or pace; 5=Severe akathisia. Strong compulsion to pace up and down most of the time. Constant restlessness associated with intense distress and insomnia. Higher scores indicated more akathisia.
Time Frame: Baseline, Week 171
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rollover Cohort: SD-809 ER | Switch Cohort: SD-809 ER
Number analyzed (Participants) | 82 | 37
units on a scale
  Baseline: number analyzed (Participants) | 78 | 37
  Baseline | 0.5 (0.83) | 0.4 (0.68)
  Change at Week 171: number analyzed (Participants) | 72 | 2
  Change at Week 171 | 0.4 (0.79) | 1.0 (1.41)

27. Secondary Outcome: Change From Baseline in Hospital Anxiety and Depression Scale (HADS) Anxiety Subscale Score at Week 171
Description: HADS is a self-administered instrument reliable for detecting states of depression and anxiety It includes 2 subscales: Hospital Anxiety and Depression Scale - anxiety (HADS-A) assesses state of generalized anxiety (anxious mood, restlessness, anxious thoughts, panic attacks); Hospital Anxiety and Depression Scale - depression (HADS-D) assesses state of lost interest and diminished pleasure response (lowering of hedonic tone). Each subscale comprised of 7 items with range 0 (no presence of anxiety or depression) to 3 (severe feeling of anxiety or depression). Total score ranged from 0 to 21 for each subscale; where higher score indicated greater severity of anxiety and depression symptoms.
Time Frame: Baseline, Week 171
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rollover Cohort: SD-809 ER | Switch Cohort: SD-809 ER
Number analyzed (Participants) | 82 | 37
units on a scale
  Baseline: number analyzed (Participants) | 79 | 37
  Baseline | 2.7 (2.99) | 4.3 (3.45)
  Change at Week 171: number analyzed (Participants) | 7 | 2
  Change at Week 171 | 1.3 (2.63) | -2.5 (2.12)

28. Secondary Outcome: Change From Baseline in Hospital Anxiety and Depression Scale (HADS) Depression Subscale Score at Week 171
Description: as for outcome 27
Time Frame: Baseline, Week 171
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rollover Cohort: SD-809 ER | Switch Cohort: SD-809 ER
Number analyzed (Participants) | 82 | 37
units on a scale
  Baseline: number analyzed (Participants) | 78 | 37
  Baseline | 2.0 (2.47) | 3.4 (2.54)
  Change at Week 171: number analyzed (Participants) | 7 | 2
  Change at Week 171 | 2.4 (5.26) | 2.0 (4.24)

29. Secondary Outcome: Change From Baseline in Epworth Sleepiness Scale (ESS) Total Score at Week 171
Description: ESS is a self-administered questionnaire comprised of 8 questions that provides a measure of a participant's general level of daytime sleepiness. Participants were asked to rate their usual chances of dozing off or falling asleep in different situations or activities that most people engage in as part of their daily lives (sitting and reading; watching TV; sitting inactive in a public place; as a passenger in a car for an hour without a break; lying down to rest in the afternoon when circumstances permit; sitting and talking to someone; sitting quietly after a lunch without alcohol; in a car, while stopped for a few minutes in traffic), on a 4-point Likert scale ranging from 0 to 3, where 0=no chance; 1=slight chance; 2=moderate chance; 3=high chance. Total ESS score is the sum of 8 item-scores and can range between 0 and 24 with a higher the score indicating a higher level of daytime sleepiness.
Time Frame: Baseline, Week 171
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rollover Cohort: SD-809 ER | Switch Cohort: SD-809 ER
Number analyzed (Participants) | 82 | 37
units on a scale
  Baseline: number analyzed (Participants) | 78 | 37
  Baseline | 4.4 (3.72) | 6.0 (4.15)
  Change at Week 171: number analyzed (Participants) | 7 | 2
  Change at Week 171 | 4.7 (7.45) | 1.0 (1.41)

30. Secondary Outcome: Number of Participants With Positive Response on the Columbia Suicide Severity Rating Scale (C-SSRS)
Description: C-SSRS is a clinician rated assessment of suicidal behavior and ideation categorized as: Suicidal behavior=a "yes" response to any of 5 suicidal behavior questions (preparatory acts or behavior, aborted attempt, interrupted attempt, non-fatal suicide attempt, and completed suicide); Suicidal ideation=a "yes" response to any one of 5 suicidal ideation questions which includes wish to be dead, non-specific active suicidal thoughts, active suicidal ideation with any methods (not plan) without intent to act, active suicidal ideation with some intent to act without specific plan, active suicidal ideation with specific plan and intent. Number of participants with positive response (response of "yes") to suicidal behavior, ideation or any non-suicidal self-injurious behavior was reported.
Time Frame: Baseline up to 1-week follow-up visit (up to approximately 3 years 9 months)
Population: as for outcome 23
Measure: Count of Participants; unit: Participants
Arm/Group | Rollover Cohort: SD-809 ER | Switch Cohort: SD-809 ER
Number analyzed (Participants) | 81 | 37
Participants
  Suicidal Ideation | 11 | 4
  Suicidal Behavior | 3 | 1
  Self-injurious behavior without suicidal intent | 1 | 0

31. Secondary Outcome: Change From Baseline in Montreal Cognitive Assessment (MoCA) Total Score at Week 171
Description: MoCA is a validated rapid screening instrument for assessing mild cognitive dysfunction. It assesses different cognitive domains: attention and concentration, executive functions, memory, language, visuoconstructional skills, conceptual thinking, calculations, and orientation by using 30 questions test. Time to administer the MoCA© is approximately 10 minutes. The total possible score ranges from 0 (worst) to 30 (best) points; where higher scores indicate better cognitive function. A score of 26 or above is considered normal and a score below 26 is considered as recognitive dysfunction.
Time Frame: Baseline, Week 171
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rollover Cohort: SD-809 ER | Switch Cohort: SD-809 ER
Number analyzed (Participants) | 82 | 37
units on a scale
  Baseline: number analyzed (Participants) | 80 | 37
  Baseline | 23.9 (4.35) | 21.9 (3.86)
  Change at Week 171: number analyzed (Participants) | 7 | 2
  Change at Week 171 | -3.1 (4.81) | 4.5 (3.54)

32. Secondary Outcome: Change From Baseline in Unified Huntington's Disease Rating Scale (UHDRS) Total Behavior Score at Week 171
Description: The UHDRS is a research tool developed by the Huntington Disease (HD) Study Group to provide a uniform assessment of the clinical features and course of HD. The components of the full UHDRS assess motor function, cognition, behaviour, functional abilities, independence scale and total functional capacities. The total behavior score is made up of subscores evaluating depressed mood, apathy, low self-esteem/guilt, compulsive behavior, anxiety, irritable behavior, perseverative/obsessive thinking, disruptive/aggressive behavior, suicidal thoughts, delusions, and hallucinations. For each subscore the frequency and severity was assessed separately. Frequency was rated on a scale of 0 (never or almost never) to 4 (very frequently, most of the time). Severity was rated on a scale of 0 (no evidence) to 4 (severe). Total behavior score ranges from 0 (no impairment) to 88 (severe impairment). Higher scores indicated greater behavioral impairments.
Time Frame: Baseline, Week 171
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rollover Cohort: SD-809 ER | Switch Cohort: SD-809 ER
Number analyzed (Participants) | 82 | 37
units on a scale
  Baseline: number analyzed (Participants) | 80 | 37
  Baseline | 7.1 (8.26) | 10.9 (10.66)
  Change at Week 171: number analyzed (Participants) | 7 | 2
  Change at Week 171 | 8.6 (12.47) | 4.5 (2.12)

33. Secondary Outcome: Change From Baseline in UHDRS Functional Assessment Score at Week 28
Description: The UHDRS is a research tool developed by HD Study Group to provide a uniform assessment of the clinical features and course of HD. The components of the full UHDRS assess motor function, cognition, behaviour, functional abilities, independence scale and total functional capacities. Functional assessment included 25 questions with possible answers 'yes' or 'no'. Total score ranges from 0 (worst) to 25 (best). Higher scores indicate better functional ability.
Time Frame: Baseline, Week 28
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rollover Cohort: SD-809 ER | Switch Cohort: SD-809 ER
Number analyzed (Participants) | 82 | 37
units on a scale
  Baseline | 21.4 (3.00) | 18.2 (4.94)
  Change at Week 28: number analyzed (Participants) | 77 | 34
  Change at Week 28 | -1.6 (2.76) | -1.6 (3.62)

34. Secondary Outcome: Change From Baseline in UHDRS Independence Scale Score at Week 28
Description: UHDRS: research tool to provide a uniform assessment of clinical features and course of HD. Components of UHDRS assess motor function, cognition, behaviour, functional abilities, independence scale and total functional capacities. Independence scale ranges from 10-100, indicating most accurate current level of participant's independence. 10=Tube fed, total bed care; 20=No speech, must be fed; 30=Participant provides minimal assistance in own feeding,bathing,toileting; 40=Chronic care facility needed; limited self-feeding; 50=24-hour supervision appropriate; assistance required for bathing,eating,toileting; 60=Needs minor assistance in dressing,toileting,bathing; 70=Self-care maintained for bathing,limited household duties; unable to manage finances; 80=Pre-disease level of employment changes or ends; cannot perform household chores, may need help with finances; 90=No physical care needed(difficult tasks avoided); 100=No special care needed. Higher scores indicate better independence.
Time Frame: Baseline, Week 28
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rollover Cohort: SD-809 ER | Switch Cohort: SD-809 ER
Number analyzed (Participants) | 82 | 37
units on a scale
  Baseline | 84.0 (9.48) | 75.5 (11.59)
  Change at Week 28: number analyzed (Participants) | 77 | 33
  Change at Week 28 | -4.2 (9.60) | -1.2 (8.93)

35. Secondary Outcome: Change From Baseline in UHDRS Total Functional Capacity (TFC) Score at Week 132
Description: UHDRS is a research tool developed by HD Study Group to provide a uniform assessment of the clinical features and course of HD. Components of the full UHDRS assess motor function, cognition, behaviour, functional abilities, independence scale and total functional capacities (TFC). TFC is a 5-item clinician rating scale typically completed after a brief interview with a participant and/or collateral source. TFC globally assesses occupation, finances, domestic chores, activities of daily living, and level of care, with scores on each item ranging from 0 to either 2 or 3 (e.g., Occupation: 0 = unable, 1 = marginal work only, 2 = reduced capacity for usual job, 3 = normal). The five items are summed to yield a TFC total score, which ranges from 0 (normal function) to 13 (severe dysfunction). Higher scores indicated better functioning.
Time Frame: Baseline, Week 132
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rollover Cohort: SD-809 ER | Switch Cohort: SD-809 ER
Number analyzed (Participants) | 82 | 37
units on a scale
  Baseline | 9.6 (2.17) | 8.3 (2.11)
  Change at Week 132: number analyzed (Participants) | 57 | 28
  Change at Week 132 | -3.1 (2.86) | -3.1 (2.71)

36. Secondary Outcome: Change From Baseline in UHDRS Cognitive Assessment Score at Week 171
Description: Components of UHDRS assess motor function,cognition,behaviour,functional abilities,independence scale, total functional capacities. Cognitive assessment component:verbal fluency(VF) score (memory,attention)(requiring participant to generate as many words as possible beginning with a specific letter[F,A,S]in 60 seconds [sec]. Score[no range]:total number of correct words for 3 letters), symbol digit modalities test(SDMT) score(psychomotor speed,attention)(participant is required to pair digits to assigned symbols using a reference key. Score[0 {worst}-120 {best}]:total number of correct written responses in 90 sec), & Stroop interference(SI) score (selective attention,executive function)(includes 3 conditions:naming colour blocks[blue, red or green]; reading colour words printed in black ink; naming ink colour of incongruous colour words. For each condition score(no range)is number of correct responses produced in 45 sec). In these tests, higher scores reflect better cognitive ability.
Time Frame: Baseline, Week 171
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rollover Cohort: SD-809 ER | Switch Cohort: SD-809 ER
Number analyzed (Participants) | 82 | 37
units on a scale
  VF Score: Baseline: number analyzed (Participants) | 80 | 37
  VF Score: Baseline | 25.1 (11.00) | 21.5 (10.79)
  VF Score: Change at Week 171: number analyzed (Participants) | 7 | 2
  VF Score: Change at Week 171 | -10.9 (10.12) | 4.0 (5.66)
  SDMT: Baseline: number analyzed (Participants) | 79 | 34
  SDMT: Baseline | 24.4 (8.91) | 22.7 (17.38)
  SDMT: Change at Week 171: number analyzed (Participants) | 7 | 2
  SDMT: Change at Week 171 | -9.6 (7.04) | 0.0 (7.07)
  SI Score: Baseline: number analyzed (Participants) | 80 | 37
  SI Score: Baseline | 3.2 (10.87) | -0.5 (6.38)
  SI Score: Change at Week 171: number analyzed (Participants) | 7 | 2
  SI Score: Change at Week 171 | -2.4 (7.42) | 6.5 (4.27)

37. Secondary Outcome: Change From Baseline in UHDRS Motor Assessment: Total Maximal Chorea (TMC) Score at Week 171
Description: UHDRS is a research tool developed by HD Study Group to provide a uniform assessment of the clinical features and course of HD. Components of the full UHDRS assess motor function, cognition, behaviour, functional abilities, independence scale and total functional capacities. Motor function assessment includes total motor score (TMS) and TMC score. TMC score is determined from Item 12 (maximal chorea) of UHDRS TMS and quantifies chorea based on assessments of the face, bucco-oral-lingual area, trunk, and the 4 extremities. TMC score is a sum of chorea scores in the 7 body regions, ranging from 0 (absent chorea) to 28 (marked/prolonged chorea). Lower TMC scores indicated less chorea.
Time Frame: Baseline, Week 171
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rollover Cohort: SD-809 ER | Switch Cohort: SD-809 ER
Number analyzed (Participants) | 82 | 37
units on a scale
  Baseline: number analyzed (Participants) | 78 | 37
  Baseline | 12.04 (4.113) | 12.46 (5.221)
  Change at Week 171: number analyzed (Participants) | 7 | 2
  Change at Week 171 | -3.71 (7.544) | 4.75 (1.061)

38. Secondary Outcome: Change From Week 8 in UHDRS Motor Assessment: TMC Score at Week 171
Description: UHDRS is a research tool developed by HD Study Group to provide a uniform assessment of clinical features and course of HD. Components of full UHDRS assess motor function, cognition, behaviour, functional abilities, independence scale and total functional capacities. Motor function assessment includes TMS and TMC score. TMC score is determined from Item 12 (maximal chorea) of UHDRS TMS and quantifies chorea based on assessments of the face, bucco-oral-lingual area, trunk, and the 4 extremities. TMC score is a sum of chorea scores in the 7 body regions, ranging from 0(absent chorea) to 28 (marked/prolonged chorea). Lower TMC scores indicated less chorea. Data was measured and available for total safety population. Data was not available by individual cohorts (rollover cohort and switch cohort) from Week 8 to Week 171, as was done for change from baseline. Therefore, in order to present results data for this outcome measure, the total, combined safety population treatment arm was used.
Time Frame: Week 8, Week 171
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Combined Cohort (Rollover and Switch): SD-809 ER: Participants of rollover cohort and switch cohort were included in this arm for the purpose of reporting data of this outcome measure.
Arm/Group | Combined Cohort (Rollover and Switch): SD-809 ER
Number analyzed (Participants) | 119
units on a scale
  Week 8: number analyzed (Participants) | 116
  Week 8 | 8.5 (4.67)
  Change at Week 171: number analyzed (Participants) | 9
  Change at Week 171 | 2.4 (5.00)

39. Secondary Outcome: Change From Baseline in UHDRS Motor Assessment: Total Motor Score (TMS) at Week 171
Description: UHDRS is a research tool developed by HD Study Group to provide a uniform assessment of the clinical features and course of HD. Components of the full UHDRS assess motor function, cognition, behaviour, functional abilities, independence scale and total functional capacities. Motor function assessment includes TMS and TMC score. The UHDRS TMS assesses all the motor features of HD and includes maximal chorea, maximal dystonia, ocular pursuit, saccade initiation and velocity, dysarthria, tongue protrusion, finger tapping, hand pronation and supination, luria, rigidity, bradykinesia, gait, tandem walking, and retropulsion pull test. Each of these was rated on a scale of 0 (normal motor function) to 4 (severely impaired motor function). TMS score is a sum of individual scores ranging from 0 (normal motor function) to 124 (severely impaired motor function). Lower TMS scores indicate better motor function.
Time Frame: Baseline, Week 171
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rollover Cohort: SD-809 ER | Switch Cohort: SD-809 ER
Number analyzed (Participants) | 82 | 37
units on a scale
  Baseline: number analyzed (Participants) | 78 | 37
  Baseline | 34.67 (16.119) | 37.76 (18.605)
  Change at Week 171: number analyzed (Participants) | 7 | 2
  Change at Week 171 | 11.29 (14.762) | 18.50 (3.536)

40. Secondary Outcome: Change From Week 8 in UHDRS Motor Assessment: TMS at Week 171
Description: Components of full UHDRS assess motor function,cognition,behaviour,functional abilities,independence scale,total functional capacities. Motor function assessment includes TMS and TMC score. TMS assesses all motor features of HD and includes maximal chorea, maximal dystonia,ocular pursuit,saccade initiation and velocity,dysarthria,tongue protrusion,finger tapping,hand pronation and supination,luria rigidity,bradykinesia,gait,tandem walking,retropulsion pull test. Each of these was rated on a scale of 0(normal motor function) to 4(severely impaired motor function). TMS score is a sum of individual scores ranging from 0(normal motor function) to 124(severely impaired motor function). Lower TMS scores= better motor function. Data was available for total safety population, not by individual cohorts(rollover and switch cohort) from Week 8 to Week 171,as was done for change from baseline. Therefore, in order to present results data,the total,combined safety population treatment arm was used.
Time Frame: Week 8, Week 171
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Combined Cohort (Rollover and Switch): SD-809 ER
Number analyzed (Participants) | 119
units on a scale
  Week 8: number analyzed (Participants) | 116
  Week 8 | 30.7 (17.40)
  Change at Week 171: number analyzed (Participants) | 9
  Change at Week 171 | 22.2 (12.02)

ADVERSE EVENTS:
Time Frame: Baseline to follow-up visit (up to approximately 3 years 9 months)
Description: Safety population included all participants who received at least 1 dose of study drug.
Arm/Group | Rollover Cohort: SD-809 ER | Switch Cohort: SD-809 ER
All-Cause Mortality (participants affected / at risk) | 1/82 | 0/37
Serious Adverse Events (participants affected / at risk) | 21/82 | 11/37
Other Adverse Events (participants affected / at risk) | 74/82 | 32/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rollover Cohort: SD-809 ER (N=82) | Switch Cohort: SD-809 ER (N=37)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 1 (1) | 0 (0)
Sudden cardiac death (General disorders) | 1 (1) | 0 (0)
Actinomycotic pulmonary infection (Infections and infestations) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis staphylococcal (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 2 (2)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection bacterial (Infections and infestations) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Penile cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Renal oncocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 1 (1)
Aggression (Psychiatric disorders) | 1 (2) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Depression suicidal (Psychiatric disorders) | 1 (1) | 0 (0)
Major depression (Psychiatric disorders) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 2 (2) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Spinal fusion surgery (Surgical and medical procedures) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rollover Cohort: SD-809 ER (N=82) | Switch Cohort: SD-809 ER (N=37)
Bradycardia (Cardiac disorders) | 0 (0) | 2 (2)
Cerumen impaction (Ear and labyrinth disorders) | 0 (0) | 2 (2)
Dry eye (Eye disorders) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 7 (7) | 5 (6)
Diarrhoea (Gastrointestinal disorders) | 11 (13) | 7 (11)
Dry mouth (Gastrointestinal disorders) | 4 (4) | 4 (4)
Dysphagia (Gastrointestinal disorders) | 7 (12) | 6 (7)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 2 (2)
Nausea (Gastrointestinal disorders) | 8 (8) | 3 (3)
Vomiting (Gastrointestinal disorders) | 7 (10) | 2 (2)
Chest pain (General disorders) | 2 (2) | 2 (2)
Fatigue (General disorders) | 7 (8) | 2 (2)
Gait disturbance (General disorders) | 4 (5) | 2 (3)
Irritability (General disorders) | 11 (13) | 4 (5)
Oedema peripheral (General disorders) | 0 (0) | 2 (2)
Pyrexia (General disorders) | 1 (1) | 2 (2)
Bronchitis (Infections and infestations) | 5 (5) | 2 (2)
Nasopharyngitis (Infections and infestations) | 8 (11) | 6 (8)
Pneumonia (Infections and infestations) | 1 (1) | 5 (5)
Sinusitis (Infections and infestations) | 3 (3) | 2 (3)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 2 (3)
Urinary tract infection (Infections and infestations) | 12 (18) | 4 (5)
Contusion (Injury, poisoning and procedural complications) | 7 (11) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 30 (78) | 15 (27)
Laceration (Injury, poisoning and procedural complications) | 7 (10) | 5 (9)
Weight decreased (Investigations) | 11 (12) | 8 (8)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 4 (5)
Dehydration (Metabolism and nutrition disorders) | 3 (3) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (5) | 2 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (2)
Akathisia (Nervous system disorders) | 5 (5) | 4 (5)
Balance disorder (Nervous system disorders) | 0 (0) | 2 (2)
Chorea (Nervous system disorders) | 7 (7) | 7 (10)
Cognitive disorder (Nervous system disorders) | 3 (4) | 2 (2)
Headache (Nervous system disorders) | 6 (7) | 1 (1)
Memory impairment (Nervous system disorders) | 3 (3) | 2 (2)
Parkinsonism (Nervous system disorders) | 3 (3) | 3 (4)
Somnolence (Nervous system disorders) | 16 (22) | 11 (16)
Agitation (Psychiatric disorders) | 3 (3) | 3 (3)
Anxiety (Psychiatric disorders) | 22 (32) | 13 (14)
Apathy (Psychiatric disorders) | 5 (6) | 1 (1)
Depressed mood (Psychiatric disorders) | 0 (0) | 2 (3)
Depression (Psychiatric disorders) | 26 (35) | 7 (8)
Insomnia (Psychiatric disorders) | 19 (23) | 6 (7)
Sleep disorder (Psychiatric disorders) | 5 (6) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 4 (6) | 2 (2)
Micturition urgency (Renal and urinary disorders) | 3 (3) | 2 (2)
Pollakiuria (Renal and urinary disorders) | 7 (7) | 1 (1)
Choking (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (4)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 3 (4) | 2 (2)
Hypotension (Vascular disorders) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.

DOCUMENTS (2):
  • Study Protocol (2015-03-02): https://cdn.clinicaltrials.gov/large-docs/96/NCT01897896/Prot_000.pdf
  • Statistical Analysis Plan (2017-09-15): https://cdn.clinicaltrials.gov/large-docs/96/NCT01897896/SAP_001.pdf